CLINICAL TRIAL: NCT06285435
Title: Activation of Coagulation as an Indicator of a Pro-thrombotic State in Patients With Pemphigus: A Case-control Study
Brief Title: Coagulation Activation in Patients With Pemphigus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Youstina Zaghloul, Master degree student, Assiut University
Other Study IDs: coagulation activation in PV
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pemphigus vulgaris patients
  Interventions: Diagnostic Test: prothrombin fragment 1+2
- control group
  Interventions: Diagnostic Test: prothrombin fragment 1+2

INTERVENTIONS:
Diagnostic Test: prothrombin fragment 1+2 — Blood sample
  Other Names: D-dimer

SUMMARY:
Aim of work:

1. To evaluate the plasma markers of coagulation activation: prothrombin F1+2 and d-dimer levels in pemphigus patients with active disease and compare them with age and sex-matched controls.
2. To evaluate the correlation of these markers with disease severity score by using Pemphigus Disease Area Index (PDAI) and with disease activity by measurement of anti-desmoglein 1 and 3 antibody titers.

DETAILED DESCRIPTION:
Pemphigus encompasses a group of autoimmune bullous diseases characterized clinically by the presence of flaccid blisters and erosions of the mucous membranes and/or skin. It is characterized by autoantibodies directed against the desmosomal desmogleins; Desmoglein 1 (Dsg1) and Desmoglein 3 (Dsg3) on keratinocyte cell surfaces resulting in acantholysis, which is the mechanism underlying pemphigus.

Pemphigus diseases can be classified into 4 main forms based on clinical and immunopathological features: pemphigus vulgaris, in about 70-80% of patients; pemphigus foliaceus, in about 20%; paraneoplastic pemphigus, in about 5%; and IgA pemphigus, in 1-3%.

The global incidence of PV ranges from 0.7 to 5 cases per million per year. PV predominantly affects adults in the 4th-6th decade of life. PV often begins with painful, non-healing erosions in oral mucosa, and develops into blisters in the skin.

The diagnosis of pemphigus is based on triad of history taking, clinical examination and immunologic investigations. ELISA using recombinant Dsgs enables detection of circulating autoantibodies in pemphigus. The sensitivity and specificity of anti-Dsg ELISA are 96% to 100% .The autoantibody titers often fluctuate in parallel with disease activity and decline with clinical improvement; therefore, these titers are useful not only for diagnosis but also for monitoring of disease activity and a decrease in the ELISA index value can be a useful guide for steroid tapering in the lesion-free phase.

Growing evidence has suggested that several autoimmune disorders are significantly associated with an increased risk of venous thromboembolism (VTE). However, the primary contribution of pemphigus to VTE development is unclear.

A retrospective cohort study demonstrated a 5% venous thromboembolism rate in patients with pemphigus within the first year after diagnosis.

A large-scale population-based longitudinal cohort study concluded that pemphigus is associated with an increased risk of pulmonary embolism (PE), particularly during the 1st year of the disease.

The mechanism underlying the increased VTE risk in pemphigus had not been clearly defined. However, there is evidence that systemic inflammation, which exists in pemphigus as well as in other autoimmune diseases, may promote thrombosis through upregulation of pro-coagulation systems, anticoagulant suppression, and antifibrinolytic effects. Elevated levels of tumor necrosis alpha (TNF-α) and interleukin (IL)-1, IL-6 and IL-8 released into systemic circulation have been found to promote coagulation.

Additional possible risk factors for VTE development in patients with pemphigus are hospitalization, immobility and high prevalence of infections. Corticosteroid therapy, the mainstay of pemphigus treatment, increases the risk of VTE by increasing the levels of fibrinogen and clotting factors.

D-Dimer is a biomarker of fibrin formation and degradation. So far, the guidelines for the diagnosis and treatment of PE have clearly stated that only D-dimer tests are used in laboratory tests for diagnosis to date.

Although D-dimer is considered a sensitive biomarker for thromboembolic events, it does not show as much specificity. Other conditions can also raise D-dimer level, such as pregnancy, renal failure and sepsis. An elevated D-dimer value is not sufficient to establish the diagnosis of pulmonary thromboembolism.

The most important marker of coagulation activation is the prothrombin fragment 1 + 2 (F1 + 2), which is a small peptide released when prothrombin is converted to thrombin by the prothrombinase complex on negatively charged phospholipids expressed on membranes of activated platelets. Consequently, an increased rate of conversion of prothrombin to thrombin, as it may occur in prothrombotic states, should result in an increase of F1 + 2 concentration in plasma. Owing to its relatively short half-life (approximately 90 minutes), the plasma levels of F1 + 2 are considered as reliable estimates of thrombin formation in vivo at the time of blood sampling.

ELIGIBILITY:
Inclusion Criteria:

* pemphigus vulgaris patients at active stage of the disease.
* patients between the ages of 18 and 60.

Exclusion Criteria:

* Patients with other autoimmune bullous diseases.
* Patients with other skin diseases.
* Patients with chronic liver, renal or haematological diseases.
* Patients with malignant tumors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with active pemphigus who are either in a relapse for less than a week or are newly diagnosed cases will be included. The active stage of PV is defined as the de novo development of blisters on a healthy (unaffected or healed) site of either the skin or the mucous membrane.
  Clinical assessment, histopathological analysis (acantholysis and intraepidermal splitting) will be used to confirm the diagnosis of each patient.
  Control group: Healthy age and sex-matched subjects, who are free of chronic systemic diseases or dermatological conditions, will be enrolled as control.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of coagulation activation markers in pemphigus patients with controls | Baseline
  Evaluate the plasma markers of coagulation activation: prothrombin F1+2 and d-dimer levels in pemphigus patients with active disease and compare them with age and sex-matched controls.

SECONDARY OUTCOMES:
Correlation of markers with disease severity | Baseline
  Evaluate correlation of these markers with disease severity score by using Pemphigus Disease Area Index (PDAI) and with disease activity by measurement of anti-desmoglein 1 and 3 antibody titers.

REFERENCES:
- [Result] Gregoriou S, Efthymiou O, Stefanaki C, Rigopoulos D. Management of pemphigus vulgaris: challenges and solutions. Clin Cosmet Investig Dermatol. 2015 Oct 21;8:521-7. doi: 10.2147/CCID.S75908. eCollection 2015. PMID 26543381
- [Result] Jiang C, Adjei S, Santiago S, Lu J, Duran M, Tyring S. Novel use of dupilumab in pemphigus vulgaris and pemphigus foliaceus. JAAD Case Rep. 2023 Sep 30;42:12-15. doi: 10.1016/j.jdcr.2023.09.018. eCollection 2023 Dec. No abstract available. PMID 37965194
- [Result] Beek NV, Zillikens D, Schmidt E. Bullous Autoimmune Dermatoses-Clinical Features, Diagnostic Evaluation, and Treatment Options. Dtsch Arztebl Int. 2021 Jun 18;118(24):413-420. doi: 10.3238/arztebl.m2021.0136. PMID 34369370
- [Result] Yuan Q, Yang W, Zhang X. Immune cells in pemphigus vulgaris and bullous Pemphigoid: From pathogenic roles to targeting therapies. Int Immunopharmacol. 2023 Oct;123:110694. doi: 10.1016/j.intimp.2023.110694. Epub 2023 Jul 29. PMID 37523970
- [Result] Kridin K, Kridin M, Amber KT, Shalom G, Comaneshter D, Batat E, Cohen AD. The Risk of Pulmonary Embolism in Patients With Pemphigus: A Population-Based Large-Scale Longitudinal Study. Front Immunol. 2019 Jul 24;10:1559. doi: 10.3389/fimmu.2019.01559. eCollection 2019. PMID 31396203
- [Result] Shaheen MS, Silverberg JI. Association of inflammatory skin diseases with venous thromboembolism in US adults. Arch Dermatol Res. 2021 May;313(4):281-289. doi: 10.1007/s00403-020-02099-6. Epub 2020 Jul 8. PMID 32642810
- [Result] Yang P, Li H, Zhang J, Xu X. Research progress on biomarkers of pulmonary embolism. Clin Respir J. 2021 Oct;15(10):1046-1055. doi: 10.1111/crj.13414. Epub 2021 Aug 3. PMID 34214256
- [Result] Marin M, Orso D, Federici N, Vetrugno L, Bove T. D-dimer specificity and clinical context: an old unlearned story. Crit Care. 2021 Mar 10;25(1):101. doi: 10.1186/s13054-021-03532-6. No abstract available. PMID 33691711
- [Result] Capecchi M, Scalambrino E, Griffini S, Grovetti E, Clerici M, Merati G, Chantarangkul V, Cugno M, Peyvandi F, Tripodi A. Relationship between thrombin generation parameters and prothrombin fragment 1 + 2 plasma levels. Int J Lab Hematol. 2021 Oct;43(5):e248-e251. doi: 10.1111/ijlh.13462. Epub 2021 Jan 12. No abstract available. PMID 33433957
- [Result] Lee SH, Hong WJ, Kim SC. Analysis of Serum Cytokine Profile in Pemphigus. Ann Dermatol. 2017 Aug;29(4):438-445. doi: 10.5021/ad.2017.29.4.438. Epub 2017 Jun 21. PMID 28761292
- [Result] Rosenbach M, Murrell DF, Bystryn JC, Dulay S, Dick S, Fakharzadeh S, Hall R, Korman NJ, Lin J, Okawa J, Pandya AG, Payne AS, Rose M, Rubenstein D, Woodley D, Vittorio C, Werth BB, Williams EA, Taylor L, Troxel AB, Werth VP. Reliability and convergent validity of two outcome instruments for pemphigus. J Invest Dermatol. 2009 Oct;129(10):2404-10. doi: 10.1038/jid.2009.72. Epub 2009 Apr 9. PMID 19357707
- [Result] Leshem YA, Atzmony L, Dudkiewicz I, Hodak E, Mimouni D. Venous thromboembolism in patients with pemphigus: A cohort study. J Am Acad Dermatol. 2017 Aug;77(2):256-260. doi: 10.1016/j.jaad.2017.01.059. Epub 2017 May 9. PMID 28495498
- [Result] Egami S, Yamagami J, Amagai M. Autoimmune bullous skin diseases, pemphigus and pemphigoid. J Allergy Clin Immunol. 2020 Apr;145(4):1031-1047. doi: 10.1016/j.jaci.2020.02.013. PMID 32272980